CLINICAL TRIAL: NCT04852289
Title: A Clinical Observational Study of SARS-CoV-2 Specific CD8 T-Cell Responses to COVID-19 Vaccines in Humans
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000383; 000383-AG
Record Dates: First submitted 2021-04-20; First posted 2021-04-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12-17

CONDITIONS: COVID-19
Keywords: Longevity; Cellular Immune; Antibodies; Natural History
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- >=65 Female: Older Females
- >=65 Male: Older Males
- 18-64 Female: Young Females
- 18-64 Male: Young Males

SUMMARY:
Background:

The immune response is how the body recognizes and defends itself against foreign and harmful substances. Researchers want to compare the immune responses between young and older healthy adults after they receive vaccine doses for COVID-19. This research may help to determine whether age impacts cell response to COVID-19 vaccines.

Objective:

To study the immune response of people who receive Pizer or Moderna COVID-19 vaccines.

Eligibility:

People aged 18 and older who have not had COVID-19 and who either plan to receive the first dose of a COVID-19 vaccine within the next month or have received at least the first of 2 doses of the vaccine within the last 6 months.

Design:

Participants will be screened by telephone.

Participants will not get the COVID-19 vaccine in this study. They must get it through a vaccine location.

Participants who have not yet been vaccinated will have 7 visits. The first 4 visits will occur in the first month before and after each vaccination. The last 3 visits will occur 6 months, 1 year, and 2 years after completed vaccination.

Participants who have received at least 1 of 2 doses of the COVID-19 vaccine within the last 6 months will have 3 visits. The first visit will occur within 6 months of receiving the first vaccine dose. The last 2 visits will occur 1 year and 2 years after the first vaccine dose.

At visits, participant will review their medical history. Their height, weight, and/or vital signs will be measured. They will give blood samples after fasting. They may give urine samples. They may have a nasal swab test for COVID-19.

DETAILED DESCRIPTION:
Study Description:

This study is to identify SARS-CoV-2 S protein specific CD8 T cells in the blood of COVID-19 vaccinated participants. Pfizer and Moderna made vaccines will be used in this study. As both vaccines are mRNA-based encoding S protein of SARS-CoV-2 and require two doses, the CD8 T cell response is expected to be comparable. We will also measure general health factors using blood samples. By analyzing the frequency, differentiation, and expansion of these SARS-CoV-2 S protein specific CD8 T cells, we hope to shed light into the CD8 T cell response to COVID-19 vaccine and its change with age.

Objectives:

To determine the proportion of individuals who develop and maintain SARS-CoV-2 S protein specific CD8 T cells after vaccination as a proxy for cellular immunity to future SARS CoV-2 exposure, to determine if there are differences in CD8 T cell response to COVID-19 vaccines between young and older healthy adults, and the longevity of CD8 T cell response over a five year follow up.

Endpoints:

Primary Endpoint: Presence or absence of various SARS-CoV-2 S protein specific CD8 T cells in COVID-19 vaccine participants and their quantitative changes during and after the course of vaccination, and over a five year time.

Secondary Endpoint: Determining the effect of age (either prespecify age >65 vs <65 or explore as a continuous variable) and sex on presence of SARS-CoV-2 S protein specific CD8 T cells

Exploratory Endpoints:

1. Correlations between CD8 T cell responses in vitro and circulating SARS-CoV-2 specific antibodies
2. Plasma inflammatory cytokines and other biomarkers

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Ability of subject to understand the study and stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female aged 18 years or older.
* Able to speak and read English.
* Willingness and ability to come to the NIH/National Institute on Aging Clinical Research Unit at MedStar Harbor Hospital or the NIH/NIA/Biomedical Research Center at Johns Hopkins Bayview campus in Baltimore for study procedures.
* No knowledge of having had SARS-CoV-2, the virus that causes COVID-19.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in

this study:

* Unable to verify identification of volunteer by state issued ID card, driver s license, or military ID. Participants earning greater than $600.00/year are issued a 1099 form, therefore, positive identification is required.
* Unable to provide informed consent.
* Current use of steroids, immunosuppressive medications, radiation therapy, or chemotherapy medications.
* Pregnancy.

In addition, eligible participants may not be immediately able to participate in the study but might be eligible at a later date. These include:

* Symptoms of a viral infection on visit 1 (defer until resolved).
* Medication: Volunteers taking the following medications would be deferred for 2 weeks after course has been completed and volunteer is feeling well: Antibiotics, antifungals, antimalarials, antivirals.
* Temporary steroids (tapers): Deferred for 72 hours after symptoms are resolved and prescription is completed if taken orally, intravenously, or intramuscular. No deferral if taken intranasal, inhaled, or for joint injection.
* Infection or Fever: Deferred until 2 weeks after antibiotics are completed and /or volunteer is feeling well.
* We wish to only select healthy confirmed COVID-19 negative patients. Therefore, those who may have a household member (co-habitant) who is newly diagnosed with COVID-19 or who has symptoms will be deferred for 14 days.
* Treatment with another investigational drug or other intervention within 14 days of visit 1 per the discretion of the Principal Investigator.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will consist of healthy men and women over 18 years of age who plan to have a COVID-19 vaccination within 30 days. An accrual ceiling of 160 participants will be recruited and screened until 140 eligible participants are enrolled, which are calculated based on four groups: young females (18-64), young males (18-64), old females (>=65), old males (>=65). Each group with 35 people to account for HLA-A2+, variations in HLA-A2 genotype percentage, and possible dropout. We will include both genders, 18 years of age and older, all races, and residents of the state of Maryland.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
We are investigating the presence or absence of various SARS-CoV-2 specific CD8 T cells in healthy COVID-19 vaccinated participants to understand the composition of CD8 T cell immunity in COVID-19 pathogenesis. | 4 months and one year data
  To determine quantitative changes of S protein specific CD8 T cells prior and post COVID-19 vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Nan-Ping P Weng, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (2):
- United States (2):
  - National Institute of Aging, Clinical Research Unit, Baltimore, Maryland
  - NIH/NIA/Biomedical Research Center at Johns Hopkins Bayview campus, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Undecided
We will deposit the research data to NCBI without individual identity information when the findings are written for publications.